CLINICAL TRIAL: NCT07091747
Title: Use of a Product Containing the Cannabinoids CBD and THC as a Treatment Strategy for Alzheimer's Disease - Alzheimer's Disease and Cannabis Clinical Trial (DAZACANN) Open-Label Phase
Acronym: DAZA OPEN
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Federal University of Latin American Integration (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, FRANCISNEY PINTO DO NASCIMENTO, University Professor, Federal University of Latin American Integration
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAZACANN Open-Label Phase; CAAE: 86640925.4.0000.8527 (Registry Identifier: BRAZIL PLATFORM)
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Alzheimer Disease (AD)
Keywords: Alzheimer's Disease; Cannabidiol (CBD); Tetrahydrocannabinol (THC); Open Label
MeSH Terms: conditions — Alzheimer Disease | interventions — nabiximols; Dronabinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open label group (Experimental): They will use the extract at a daily dose of 50 mg of CBD and 5 mg of THC from a product with a CBD:THC concentration of 50 mg/ml:5 mg/ml for a period of 24 months.
  Interventions: Other: Cannabis 50 mg of CBD and 5 mg of THC

INTERVENTIONS:
Other: Cannabis 50 mg of CBD and 5 mg of THC — Cannabis 50 mg of CBD and 5 mg of THC

SUMMARY:
Alzheimer's Disease (AD) has become a significant public health issue due to the increase in its incidence from 2.0 to 16.8 cases per thousand people in a year, based on 2022 data. As many countries experience population aging, there is an increase in the prevalence of AD cases, which is the main form of dementia in the elderly. It commonly begins around the age of 60, with aging being the primary risk factor. AD is a neurodegenerative disorder characterized by the presence of extracellular beta-amyloid plaques and intracellular neurofibrillary tangles of Tau protein. Among the main symptoms of AD is progressive memory loss, with varying degrees of cognitive impairment. These symptoms share common clinical features such as a progressive decline in cognitive functions, including abstract thinking, judgment, language, personality changes, and behavioral symptoms, as well as the emergence of certain comorbidities.

As there are currently no curative treatments for this disease, pharmacotherapy aims to control the progressive symptoms, improving cognitive and functional aspects in patients, and consequently their quality of life. In this context, there is a need for further research to identify effective drugs that can delay or alleviate symptoms.

This study is part of the second phase of the project entitled: Use of a Product Containing the Cannabinoids CBD and THC as a Treatment Strategy for Alzheimer's Disease - Alzheimer's Disease and Cannabis Clinical Trial (DAZACANN): A randomized, double-blind, placebo-controlled clinical trial previously approved by the Human Ethics Committee - CEP (CAAE 60167722.6.0000.0107). The trial is being finalized at the Laboratory of Medicinal Cannabis and Psychedelic Science, located in the city of Foz do Iguaçu, Paraná, and will continue with a new experimental design, now as an open-label trial (all participants will receive the extract and will be informed about the formulation they are receiving).

The objective of this study remains to evaluate the clinical and biochemical effects of using cannabinoid-based products with low doses of purified CBD and THC, both individually and in combination, in patients with AD.

ELIGIBILITY:
Inclusion Criteria:

* Have participated in and completed all assessments conducted in the first phase of the project.
* Agree to and sign a new informed consent form.

Exclusion Criteria:

* Patients who did not participate in the first stage.
* Patients who began participating in the first stage but withdrew at any time.
* Patients who do not agree and/or fail to sign the new informed consent form

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2025-04-07 (Actual); Primary Completion 2025-12-12 (Estimated); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
Mini Mental State Examination | 24 months
  Assess cognitive function and disease progression. Cognitive function preserved (27 to 30 points), Mild cognitive impairment (21 to 26 points), Moderate cognitive impairment (10 to 20 points), Severe cognitive impairment (0 to 9 points).

SECONDARY OUTCOMES:
Neuropsychiatric Inventory | 24 months
  Identify neuropsychiatric symptoms across different domains using the Neuropsychiatric Inventory. Score Range: 0-20 Mild symptoms or no significant impairment, 21-50 Moderate symptoms, 51-120 Severe symptoms with major impact
Quality of Life in Alzheimer's Disease scale (QoL-AD) | 24 month
  The scale has 3 versions, one of which is applied to the patient, another to the caregiver to answer about the patient's life, and one for the caregiver to answer about their own life. The score may vary, the one the investigators will use is the sum of the questionnaires about the patient, caregiver version and patient version, with the patient version having a weight of 2. Its score varies from 13, indicating the worst possible quality of life, up to 52, and the higher the score, the higher the quality of life.
Epworth Sleepiness Scale (ESS ) | 24 month
  Evaluates 8 items with scores ranging from 0 to 24, in which scores higher than 10 indicate sleep disturbances.
Specific markers of Alzheimer's disease | 24 month
  The following proteins will be quantified in the cerebrospinal fluid: beta-amyloid 40, beta-amyloid 42, tau protein (fraction 181), and phosphorylated tau protein.
Brain Derived Neurotrophic Factor | 24 month
  It will be measured in serum or plasma
Inflammatory markers | 24 month
  TNFα (Tumor Necrosis Factor alpha), IL-6 (Interleukin-6), IL-1β (Interleukin-1 beta), and IL-10 (Interleukin-10), it will be measured in serum or plasma.
Safety Endpoints - UKU Side Effect Rating Scale | 24 month
  Will be conducted on patients and caregivers during all planned visits to ascertain the frequency and severity of adverse events. There will be neurological and physical examinations as well as laboratory testing. Total Score Sum of all 48 item scores (minimum 0; maximum 144), indicates greater overall severity of psychotropic side effects.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal da Integração Latino-Americana, Foz do Iguaçu, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No